CLINICAL TRIAL: NCT04880356
Title: Clinical, Instrumental and Laboratory Data Collection of Subjects with Ultra-rare Inherited Metabolic and Degenerative Neurological Diseases
Brief Title: Longitudinal Study of Ultra-rare Inherited Metabolic and Degenerative Neurological Diseases.
Status: Recruiting | Type: Observational
Sponsor: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Responsible Party: Sponsor
Other Study IDs: MaNeNeND
Record Dates: First submitted 2021-04-19; First posted 2021-05-10 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Inherited Disease; Rare Diseases; Metabolic Disease; Undiagnosed Disease; Neurologic Disorder; Neuro-Degenerative Disease
Keywords: Leukodystrophies,; Adrenoleukodystrophy,; Metachromatic leukodystrophy,; Krabbe disease,; Vanishing White Matter Syndrome,; Alexander disease,; Hereditary Leukodystrophy with Spheroids (CSF1R-related HLDS),; Nasu-Hakola disease (TREM2- and TYROBP-related disease); Leukoencephalopathy, progressive, with ovarian failure (LKENP, AARS2-related),; Pelizaeus-Merzbacher disease,; Pelizaeus-Merzbacher-like disease,; Hypomyelinating leukodystrophies,; Leukodystrophies with calcifications and cysts (LCC),; Leukoencephalopathy with ataxia disease (LKPAT, CLCN2-related),; L-2-Hydroxyglutaric aciduria,; Polyglucosan bodies disease,; Methylmalonic acidemia with homocystinuria,; Niemann-pick type C,; Fahr's disease,; Wilson's disease,; Cerebrotendinous Xanthomatosis,; Sphingolipidoses
MeSH Terms: conditions — Genetic Diseases, Inborn; Rare Diseases; Metabolic Diseases; Undiagnosed Diseases; Nervous System Diseases; Adrenoleukodystrophy; Leukodystrophy, Metachromatic; Leukodystrophy, Globoid Cell; Alexander Disease; Polycystic lipomembranous osteodysplasia with sclerosing leukoencephalopathy; Leukoencephalopathies; Pelizaeus-Merzbacher Disease; Cysts; 2-Hydroxyglutaricaciduria; Methylmalonic acidemia with homocystinuria; Fahr's disease; Hepatolenticular Degeneration; Xanthomatosis, Cerebrotendinous; Sphingolipidoses

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Retrospective study: collection of retrospective data from adult patients with ultra-rare inherited neurological diseases
  Interventions: Other: collection of data
- Prospective study: prospective data will be collected starting from March 2021 (date of protocol approval) and spanning the next ten years
  Interventions: Other: collection of data

INTERVENTIONS:
Other: collection of data — collection of retrospective and prospective data from adult patients with ultra-rare inherited neurological diseases

SUMMARY:
General aim of the study is the improvement of the clinical knowledge of ultra-rare inherited metabolic and degenerative neurological diseases (prevalence less than 5:100,000) in adulthood through the systematic longitudinal collection of clinical, laboratory and instrumental data.

DETAILED DESCRIPTION:
The study provides a collection of retrospective data from adult patients with ultra-rare inherited neurological diseases followed at "Carlo Besta" Neurological Institute from 1st January 2004 until March 2021. Further, prospective data will be collected starting from March 2021 (date of protocol approval) and spanning the next ten years. Normal clinical practice will be followed for collection of the prospective data. Follow-up assessment will be performed at least once a year to evaluate the disease course. Based on their clinical manifestations, patients will be assessed by using quantitative functional tests (clinimetric tests such as Timed Up and Go Test) and traditional ordinal scales (such as the scale for the assessment and rating of ataxia (SARA). Moreover, a varying of laboratory and instrumental tests (e.g., neuroimaging, neurophysiological investigations, etc.) will be used according to clinical practice in selected patients.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Subjects with ultra-rare inherited degenerative and metabolic neurological diseases
* Subjects with undiagnosed neurological diseases (when supposed to be inherited)

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with ultra-rare inherited degenerative and metabolic neurological diseases
  Adults with undiagnosed neurological diseases (when supposed to be inherited)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2031-03 (Estimated); Study Completion 2031-03 (Estimated)

PRIMARY OUTCOMES:
Verbal (letter) fluency | 10 years
  Repeated Montreal Cognitive Assessment (MoCA) letter F fluency subtest
Stance and gait performances [Time Frame: 10 years] Stance and gait performances | 10 years
  Repeated SARA (Scale for the Assessment and Rating Ataxia) stance subtask, ambulation index (AI) and Timed Up and Go (TUG) test
Upper limb motor function | 10 years
  Repeated ONLS (Overall Neuropathy Limitation Scale) arm scale
Swallowing function (dysphagia) | 10 years
  Repeated NP-C mDRS (Niemann-Pick type C modified disability rating scale) swallowing scale
Speech function (dysarthria) | 10 years
  Repeated NP-C mDRS language scale
Bladder function | 10 years
  Repeated AADS (Adult Adrenoleukodystrophy Disability Score) Bladder function scale
Sleep | 10 years
  Repeated assessment of presence or absence of sleep disturbances
Quality of life | 10 years
  Repeated EuroQol-5D-5L (EQ-5D-5L) questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan, Milano, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Benzoni C, Moscatelli M, Lanteri P, Pensato V, Calo C, Allievi S, Gellera C, Ardissone A, Moroni I, Fenu S, Cavalca E, Pareyson D, Salsano E. Adrenoleukodystrophy in adults: phenotypic characterisation and natural history in a large cohort. J Neurol Neurosurg Psychiatry. 2026 Feb 10:jnnp-2025-337540. doi: 10.1136/jnnp-2025-337540. Online ahead of print. PMID 41667276
- [Derived] Moscatelli M, Benzoni C, Doniselli FM, Verri M, Pascuzzo R, Aquino D, Mazzi F, Erbetta A, Salsano E. Interval between contrast administration and T1-weighted MRI for cerebral adrenoleukodystrophy: a single-case observation. Eur Radiol Exp. 2023 Oct 2;7(1):57. doi: 10.1186/s41747-023-00373-6. PMID 37782421